CLINICAL TRIAL: NCT06808594
Title: The Use of APSI: Long Term Follow-up
Brief Title: The Use of Adaptive Proximal Scaphoid Implant (APSI): Long Term Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Massimo Corain, Director, Head of Hand Surgery Unit, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: prog.74 CET prot.67418
Record Dates: First submitted 2025-01-11; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Scaphoid Non-union Advanced Collapse (SNAC Wrist)
Keywords: osteoarthritis; arthroplasty; Scaphoid fracture; Pyrocarbon; Bone implant
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Retrospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Long term follow-up of patients treated with APSI (Experimental): Long-term clinical and radiographic outcomes in patients undergoing APSI (Adaptive Proximal Scaphoid Implant); evaluation of wrist strength and ROM (Range of Motion) on the operated side compared with the healthy side; evaluation of daily, work and sports autonomy with DASH (Disabilities of the Arm, Shoulder, and Hand) and PRWE (Patient Rated Wrist Evaluation) questionnaires and evaluating the return to normal daily, work and sports activities pre-surgery; quantification of pain at the site of surgery.
  Interventions: Device: APSI prosthesis implant

INTERVENTIONS:
Device: APSI prosthesis implant — The adaptative proximal scaphoid implant (APSI) is a pyrocarbon partial scaphoid prosthesis, ovoid and unfixed, which replaces the proximal pole of the scaphoid and allows adaptative mobility in the movements of the first chain and restores the geometry of the carpus, thus preventing the evolution in SNAC (Scaphoid Non-union Advanced Collapse). Pyrocarbon has good compatibility with joint cartilage and bone, a modulus of elasticity similar to bone minimizing stress shielding effects and resorption. The implant is designed with two radii of curvature: in the frontal plane, the smaller radius of curvature corresponds to the scaphoid fossa, and the larger radius of curvature is directed anteroposteriorly to the transverse plane. When it's correctly positioned, the smallest radius of the curvature is visible in the anteroposterior view, whereas it's greater in the lateral view. These two axes of the implant make it adaptable to the kinematics of the wrist.

SUMMARY:
Scaphoid proximal pole fracture with avascular necrosis is a complex surgical problem. In some cases, it's possible to perform a scaphoid hemiarthroplasty with an adaptative proximal scaphoid implant (APSI), made of pyrocarbon, replacing the necrotic proximal pole. APSI allows an early mobilization of the wrist, an optimal recovery of strength and a rapid return to normal daily and work activities without limitations. This implant delays palliative and more invasive surgical treatments in patients that are generally young with high functional demands. The investigators have performed a long-term follow up (with a mean follow-up of 17 years) of the early cases of APSI implant performed, starting from 1999. Radiographic and clinical strength recovery, along with subjective outcomes, have been shown to be good, with a rapid return to daily and work activities, indicating that APSI implants are a good alternative to traditional and invasive techniques.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent APSI implant surgery in the period from December 1999 to December 2016, with surgery performed via dorsal or volar approach in the case of previous surgical access;
* collection of informed consent to the processing of personal data by the Patients contacted in order to be included in the study.

Exclusion Criteria:

* patients for whom it was not possible to obtain informed consent to the processing of personal data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1999-12-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Radiographic outcome | Through study completion, an average of 17 year
  X-Rays showed that all the implants were correctly positioned, without any particular or evident erosion of the surrounding bone structures. A pattern of moderate or non-severe degree of arthrosis of the wrist could generally be found. By comparing the X-rays taken at the follow-up, it was possible to detect a general slight evolution of the arthritic in the wrist compared to what was visible at the beginning of the treatment, in all the patients.

SECONDARY OUTCOMES:
DASH (Disabilities of the Arm, Shoulder, and Hand) | Through study completion, an average of 17 year
  The DASH is a self-administered questionnaire of over 30 questions designed to measure function and symptoms in patients with any musculoskeletal disorder of the upper limb. MAX 100, MIN 0
PRWE (Patient Rated Wrist Evaluation) | Through study completion, an average of 17 year
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. MAX 50, MIN 0
VAS (Visual Analogue Scale) | Through study completion, an average of 17 year
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. MAX 10, MIN 0

IPD SHARING:
Plan to Share IPD: Yes
Database of evaluated patients